CLINICAL TRIAL: NCT00912158
Title: CPAP Versus BiPAP in Acute Cardiogenic Pulmonary Edema: Experience With 129 Patients
Brief Title: Non Invasive Mechanical Ventilation in Acute Cardiogenic Pulmonary Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Prof. Gamal R Agmy, Faculty of Medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RICU, Assiut University 1
Record Dates: First submitted 2009-04-08; First posted 2009-06-03 (Estimated); Results first posted 2009-06-03 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-08

CONDITIONS: Acute Cardiogenic Pulmonary Edema
Keywords: CPE; CPAP; BiPAP; non invasive mechanical ventilation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CPAP + ST (Active Comparator): Continuous positive airway pressure (CPAP) and Standard medical therapy (ST)
  Interventions: Device: CPAP
- BiPAP + ST (Active Comparator): Bilevel positive airway pressure (BiPAP) and standard medical therapy (ST)
  Interventions: Device: BIPAP
- ST (Active Comparator): Standard Medical therapy (ST)
  Interventions: Other: standard therapy (ST)

INTERVENTIONS:
Other: standard therapy (ST) — standard medical therapy
  Other Names: Medical treatment of acute cardiogenic pulmonary oedema
  Arms: ST
Device: CPAP — Non-invasive mechanical ventilation (CPAP)
  Other Names: Continuous postive air way pressure; noninvasive positive support ventilation (NPSV)
  Arms: CPAP + ST
Device: BIPAP — Non-invasive mechanical ventilation (BIPAP)
  Other Names: Bilevel Positive Airway Pressure ventilation
  Arms: BiPAP + ST

SUMMARY:
Cardiogenic pulmonary edema (CPE) is a common medical emergency and noninvasive ventilation (NIV) in addition to conventional medical treatment might be beneficial for patients with CPE.

DETAILED DESCRIPTION:
To evaluate the effect of adding continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP) to standard medical therapy (ST) on intensive care unit (ICU) stay, hospital stay, mortality, need for endotracheal intubation, partial arterial O2 tension (PaO2), intrapulmonary shunt, alveolar-arterial (A-a) oxygen gradient, and cardiac output in patients admitted to the respiratory intensive care unit (ICU) or cardiac care unit (CCU) with acute CPE with gas exchange abnormalities and to evaluate the impact of heart failure type on the outcome of different therapeutic schedules.

ELIGIBILITY:
Inclusion Criteria:

1. CPE confirmed radiologically and/or clinically
2. Severe acute respiratory failure (partial arterial oxygen (PaO2)/Fraction of inspired oxygen (FIO2) less than 250)
3. Dyspnea of sudden onset with respiratory
4. Systolic blood pressure < 180 mmHg

Exclusion Criteria:

1. Immediate need for endotracheal intubation:

   * Severe sensorial impairment
   * Shock
   * Ventricular arrhythmias,
   * Life-threatening hypoxia (SpO2 [oxygen saturation as indicated by pulse oximetry] less than 80% with oxygen)
   * Acute myocardial infarction necessitating thrombolysis
   * Cardiac or respiratory arrest
2. Severe chronic renal failure
3. Pneumothorax.
4. Contraindication of non invasive ventilation (NIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2003-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gamal M Agmy, MD, FCCP, Principal Investigator — Chest Department, Faculty of Medicine-Assiut University; Maha K Ghanem, MD, Study Chair — Chest Department, Faculty of Medicine- Assiut University; Hoda A Makhlouf, MD, Study Chair — Chest Department, Faculty of Medicine- Assiut University; Amany O Mohamed, MD, Study Chair — Chest Department, Faculty of Medicine- Assiut University; Hamdy S Mohamed, MD, Study Chair — Cardiology Department, Faculty of Medicine- Assiut University; Hatem A Helmy, MD, Study Chair — Cardiology Department, Faculty of Medicine - Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Chadda K, Annane D, Hart N, Gajdos P, Raphael JC, Lofaso F. Cardiac and respiratory effects of continuous positive airway pressure and noninvasive ventilation in acute cardiac pulmonary edema. Crit Care Med. 2002 Nov;30(11):2457-61. doi: 10.1097/00003246-200211000-00009. PMID 12441754
- [Background] Gray A, Goodacre S, Newby DE, Masson M, Sampson F, Nicholl J; 3CPO Trialists. Noninvasive ventilation in acute cardiogenic pulmonary edema. N Engl J Med. 2008 Jul 10;359(2):142-51. doi: 10.1056/NEJMoa0707992. PMID 18614781
- [Background] Agarwal R, Aggarwal AN, Gupta D, Jindal SK. Non-invasive ventilation in acute cardiogenic pulmonary oedema. Postgrad Med J. 2005 Oct;81(960):637-43. doi: 10.1136/pgmj.2004.031229. PMID 16210459
- [Result] Vital FM, Saconato H, Ladeira MT, Sen A, Hawkes CA, Soares B, Burns KE, Atallah AN. Non-invasive positive pressure ventilation (CPAP or bilevel NPPV) for cardiogenic pulmonary edema. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD005351. doi: 10.1002/14651858.CD005351.pub2. PMID 18646124
- See also: Medscape: Free CME, Medical News, Full-text Journal Articles & More — http://www.medscape.com
- See also: U.S. National Library of Medicine & the National Institutes of Health — http://www.pubMed.gov
- See also: The Cochrane library: Evidence for healthcare decision-making — http://www.cochrane.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location: Respiratory and Coronary Intensive Care Units of Assiut University Hospital. Patients with acute cardiogenic pulmonary oedema (CPE)
Pre-assignment Details: All enrolled participants were assigned to one of the three studied groups.
Groups:
- CPAP+ST: Continuous positive airway pressure plus standard medical therapy
- BiPAP + ST: Bilevel positive airway pressure + standard medical therapy
- Standard Treatment: Standard medical therapy alone
Period: Overall Study
Arm/Group | CPAP+ST | BiPAP + ST | Standard Treatment
Started | 44 | 44 | 41
Completed | 44 | 44 | 41
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP+ST | BiPAP + ST | Standard Treatment | Total
Number analyzed (Participants) | 44 | 44 | 41 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 10 | 36
  >=65 years | 30 | 32 | 31 | 93
Age Continuous [Mean (Standard Deviation); unit: years] | 66 (6.9) | 68 (3.8) | 69 (5.8) | 67 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 10 | 36
  Male | 30 | 32 | 31 | 93
Region of Enrollment [Number; unit: participants]
  Egypt | 44 | 44 | 41 | 129

OUTCOME MEASURES:

1. Secondary Outcome: Arterial Blood Gases, Respiratory Rate, Blood Pressure, Cardiac Output ,Intrapulmonary Shunt, A-a Oxygen Gradient, Heart Rate, and Dyspnea Duration of Hospital and ICU Stay and Mortality
Time Frame: Hospital stay
Reporting Status: Not Posted, anticipated posting 2010-01

2. Primary Outcome: Number of Patients Who Were Intubated
Description: Number of patients who were subjected to endotracheal intubation and invasive mechanical ventilation
Time Frame: During ICU Stay
Measure: Number; unit: participants
Arm/Group | CPAP+ST | BiPAP + ST | Standard Treatment
Number analyzed (Participants) | 44 | 44 | 41
participants | 5 | 4 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes